CLINICAL TRIAL: NCT04190537
Title: PARADOX - the Incidence of Paradoxical Reactions in Pediatric Patients Premedicated with Midazolam
Acronym: PARADOX
Status: Completed | Type: Observational
Sponsor: Masaryk Hospital Usti nad Labem (Other)
Responsible Party: Principal Investigator, Petr Vojtisek, Petr Vojtisek, senior consultant of paediatric anesthesia and IC, Masaryk Hospital Usti nad Labem
Other Study IDs: 273/15
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Pharmacological Action
Keywords: Paradoxial reaction midazolam

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Summary

The premedication is one of the essential sides of pediatrics anesthesia. Midazolam is considered such as standard these days. Children may develope a paradoxical reaction to benzodiazepines which is one of the adverse effect. Its incidence is unknown. The hypothesis is, in pediatric patients undergoing general anesthesia premedicated with oral midazolam, the incidence of the paradoxical reaction is 10%. Primary Goal of the study is to find out the incidence of the paradoxical reaction in pediatric patients premedicated with oral midazolam prior to general anesthesia. Secondary goal is to find out the incidence of the paradoxical reactions in children of different age groups. For the assessment, the study uses parameters: RASS, blood pressure, heart rate, PAED, PSAS, MAS and VAS.

DETAILED DESCRIPTION:
The premedication is one of the essential sides of pediatrics anesthesia. Midazolam is considered such as standard these days. Children may develope a paradoxical reaction to benzodiazepines which is one of the adverse effect.

The paradoxical reaction is an abnormal stimulative reaction to benzodiazepines characterized by hallucination, disorientation, alteration in perception and recognition as well as the escalation of negative emotion- uncalming crying, agitation, restlessness, and hostility. Risk factors for the development of the paradoxical reaction are young age, mental illness, genetic disposition, male sex, alcohol abuse, and higher midazolam doses.

The incidence of paradoxical reaction is referred to be about 1-10%, in some specific groups even more (about 29%). The exact incidence is still not known since the accurate definition of paradoxical reaction is still missing.

Primary Goal of the study is find out the incidence of the paradoxical reaction in pediatric patients premedicated with oral midazolam prior to general anesthesia and incidence of the paradoxical reactions in children of different age groups (3 months-1 year, 1 year-3 years, 3 years-6 years, 6 years-12 years, 12 years-18 years) . The calculated file size is 500 patients. All eligible patients should be evaluated for pre-treatment, pre-anesthesia, immediately prior to anesthesia and anesthesia when RASS above -2. For purpose of the study we have determined the definition of paradoxical reaction as an increase in pulse and/or blood pressure of 20% over pre-premedication , RASS increase by one point or more and raising PEAD to 10 or more points. The paradoxical reaction criteria are met if at least two points of the definition are met. Change within 45min. after premedication.

ELIGIBILITY:
Inclusion Criteria:

age from 3 months to 18 years

* oral midazolam premedication for at least 30 minutes before rating
* patient undergoing deep sedation / general anesthesia diagnostic or surgery with RASS -4 or more

Exclusion Criteria:

- personal history of benzodiazepines using

* moderate or severe respiratory insufficiency
* myopathy, neuromuscular transmission disorders
* moderate or severe CNS disability, including brain tumors, uncontrolled convulsions
* age <3 months and> 18 years
* pregnancy

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All eligible patients should be evaluated for pre-treatment, pre-anesthesia, immediately prior to anesthesia and anesthesia when RASS above -2
Sampling Method: Non-Probability Sample
Enrollment: 749 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2021-06-16 (Actual)

PRIMARY OUTCOMES:
Incidence of the paradoxical reaction in pediatric patients premedicated with oral midazolam prior to general anesthesia. | Change within 45min. after premedication
  Investigate the incidence of paradoxical reactions after administration of midazolam in the pediatric population

CONTACTS AND LOCATIONS:
Overall Officials: Petr Vojtisek, doctor, Study Chair — Masaryk Hospital Usti nad Labem
Locations (1):
- Masaryk hospital, Ústí nad Labem, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moon YE. Paradoxical reaction to midazolam in children. Korean J Anesthesiol. 2013 Jul;65(1):2-3. doi: 10.4097/kjae.2013.65.1.2. No abstract available. PMID 23904931
- [Background] Shin YH, Kim MH, Lee JJ, Choi SJ, Gwak MS, Lee AR, Park MN, Joo HS, Choi JH. The effect of midazolam dose and age on the paradoxical midazolam reaction in Korean pediatric patients. Korean J Anesthesiol. 2013 Jul;65(1):9-13. doi: 10.4097/kjae.2013.65.1.9. Epub 2013 Jul 19. PMID 23904933
- [Background] Tobin JR. Paradoxical effects of midazolam in the very young. Anesthesiology. 2008 Jan;108(1):6-7. doi: 10.1097/01.anes.0000296717.85521.b5. No abstract available. PMID 18156876
- [Background] McKenzie WS, Rosenberg M. Paradoxical reaction following administration of a benzodiazepine. J Oral Maxillofac Surg. 2010 Dec;68(12):3034-6. doi: 10.1016/j.joms.2010.06.176. Epub 2010 Oct 14. No abstract available. PMID 20950912